CLINICAL TRIAL: NCT02601495
Title: Latent Structure of Multi-level Assessments and Predictors of Outcomes for Women in Recovery
Status: Active, not recruiting | Type: Observational
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: University of Oklahoma (Other); Rutgers University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-009
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Depression; Anxiety; Eating Disorders; Drug Use Disorders; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Depression; Anxiety Disorders; Feeding and Eating Disorders; Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Serum, Plasma, Microbiome
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women in a court diversion program: Women enrolled in the court diversion program in Tulsa, Oklahoma called Women in Recovery who report symptoms related to anxiety or depressive symptoms (Patient Health Questionnaire score ≥ 10 and/or Overall Anxiety Severity and Impairment Scale ≥ 8), problematic eating behavior(Eating Disorder Screen score ≥ 2), problems related to substance use (Drug Abuse Screening Test score > 2), or post traumatic stress disorder symptoms (PTSD Checklist score ≥ 30).
  Interventions: Behavioral: Women in a court diversion program

INTERVENTIONS:
Behavioral: Women in a court diversion program — Women in Recovery (WIR) is an intensive outpatient alternative for eligible women facing long prison sentences for non-violent, drug-related offenses in Oklahoma.

SUMMARY:
In this study the investigators will seek to improve their understanding of how positive and negative valence systems, cognition, and arousal/interoception are inter-related in disorders of trauma, mood, substance use, and eating behavior for women involved in a court diversion program in Tulsa, Oklahoma (Women in Recovery). The investigators will recruit 100 individuals and use a wide range of assessment tools, neuroimaging measures, blood and microbiome collections and behavioral tasks to complete the baseline and follow-up study visits. Upon completion, the investigators aim to have robust and reliable dimensional measures that quantify these systems and a set of assessments that should be recommended as a clinical tool to enhance outcome prediction for the clinician and assist in determining who will likely benefit from the diversion program, and to inform future revision or augmentation of the program to increase treatment effectiveness.

DETAILED DESCRIPTION:
Neuroscience has made tremendous progress in understanding the basic neural circuitry that underlies important processes such as attention, memory, and basic emotion processing. Yet, little progress has been made to utilize these insights to apply them to psychiatric populations in order to make clinically meaningful predictions. The connection between psychiatric disorders and their underlying neurobiology has been difficult to establish. The overarching theme of this study is to determine how biological and objective behavioral measures can contribute to improving assessment and treatment of women who attend a court diversion program (Women in Recovery [WIR]) that includes treatment for mental health symptoms. The investigators will use the National Institute of Mental Health (NIMH) Research Domain Criteria (RDoC) framework as a heuristic approach that integrates neuroscience and psychopathology to study the positive and negative valence systems, cognition and arousal/interoception domains. Within this framework the investigators will study a group of treatment seeking individuals with mental health conditions to determine how dysfunctions of affect, substance use, and eating behavior organize across different levels and whether these latent factors can be used to generate clinically useful prediction.

Using self-report, behavior, physiology, neural circuit, cell, molecule, and gene unit of analysis measures, the investigators propose to enroll 1000 individuals from four different cohorts over 5 years: (1) anxiety and/or depression; (2) eating problems; (3) substance use problems; and (4) healthy controls. Each individual will undergo a multi-level assessment that consists of (a) a standardized diagnostic assessment, (b) self-report questionnaires, (c) behavioral tasks, (d) physiological measurements, (e) structural and functional magnetic resonance imaging (fMRI) and EEG, (f) biomarker and microbiome assessments, (g) blood to derive induced pluripotent stem cells, (h) and genetic and epigenetic assessments. These individuals will be followed up for one year and will be re-assessed using a multi-domain assessment of functioning, which will include: (a) symptom severity and duration, (b) subjective well-being, (c) psychosocial function, (c) occupational function, (d) physical health, (e) utilization of mental health resources (treatment), and (f) compliance with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Women in Recovery (WIR) program and reporting problems with:

   1. Anxiety and/or depressive symptoms
   2. Trauma-related symptoms
   3. Problems related to substance use
   4. Problems related to eating behavior
2. Screened positive for problems in (1) as indicated by:

   1. Patient Health Questionnaire (PHQ-9) ≥ 10 and/or Overall Anxiety Severity and Impairment Scale (OASIS) ≥ 8.
   2. PTSD Checklist (PCL) ≥30
   3. Drug Abuse Screening Test (DAST-10) score > 2
   4. Eating Disorder Screen (SCOFF) score ≥ 2
3. Have a body mass index between 17 to 38 kg/m²
4. Able to provide written informed consent.
5. Have sufficient proficiency in English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

1. No telephone or easy access to telephone.
2. Has a history of unstable liver or renal insufficiency; glaucoma; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
3. A positive test for drugs of abuse, including alcohol (breath test), cocaine, marijuana, opiates, amphetamines, methamphetamines, phencyclidine, benzodiazepines, barbiturates, methadone, and oxycodone.
4. Has any of the following Diagnostic and Statistical Manual (DSM-V) disorders:

   1. Schizophrenia Spectrum and Other Psychotic Disorders
   2. Bipolar and Related Disorders
   3. Obsessive-Compulsive and Related Disorders
5. Moderate to severe traumatic brain injury or other neurocognitive disorder
6. Active suicidal ideation with intent or plan.
7. Change in the dose or prescription of a medication within the 6 weeks before enrolling in the study that could affect brain functioning
8. Prescription of a medication outside of the accepted range, as determined by the best clinical practices and current research.
9. Taking drugs that affect the fMRI hemodynamic response (e.g., methylphenidate, acetazolamide, excessive caffeine intake > 1000 mg/day)
10. MRI contraindications
11. Unwillingness or inability to complete any of the major aspects of the study protocol Non-correctable vision or hearing problems

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women enrolled in a court diversion program called Women in Recovery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Diagnosis | Baseline to 1 year
  Test the predictive effects of endophenotypes (genetic, imaging and behavioral factors) on clinical diagnosis at baseline compared to one year later using the Mini International Psychiatric Interview in patients and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Martin P. Paulus, M.D., Principal Investigator — Laureate Institute for Brain Research

REFERENCES:
- [Background] Insel T, Cuthbert B, Garvey M, Heinssen R, Pine DS, Quinn K, Sanislow C, Wang P. Research domain criteria (RDoC): toward a new classification framework for research on mental disorders. Am J Psychiatry. 2010 Jul;167(7):748-51. doi: 10.1176/appi.ajp.2010.09091379. No abstract available. PMID 20595427
- [Background] Sanislow CA, Pine DS, Quinn KJ, Kozak MJ, Garvey MA, Heinssen RK, Wang PS, Cuthbert BN. Developing constructs for psychopathology research: research domain criteria. J Abnorm Psychol. 2010 Nov;119(4):631-9. doi: 10.1037/a0020909. PMID 20939653